CLINICAL TRIAL: NCT05937074
Title: Metabolic Response to Food in Lung Cancer
Acronym: METRIC
Status: Active, not recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Justin Brown, Director, Cancer Metabolism Program, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-017
Record Dates: First submitted 2023-06-23; First posted 2023-07-10 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Weight loss (%) — Change in body weight from cancer diagnosis to study enrollment

SUMMARY:
This goal of this study is to describe how unintentional weight loss influences fasting and post-prandial metabolic flexibility in participants with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Diagnosis of non-small-cell lung cancer
* Reported weight stability or loss after cancer diagnosis
* Body mass index less than or equal to 35 kilograms per meter squared
* Ability to provide written informed consent
* Willing and able to comply with all scheduled visits, treatment plans, lab tests, and other study procedure
* Allow the collection and storage of biospecimens and data for future use

Exclusion Criteria:

* Prior diagnosis of diabetes mellitus (type 1 or type 2)
* Currently pregnant or breastfeeding
* Contraindication to consuming the liquid mixed meal
* Any medications affecting gastric motility
* Any other condition that, in the investigator's opinion, would preclude participation or successful compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants with non-small-cell lung cancer with varying degrees of weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory quotient | Difference between pre- to post-prandial conditions over four hours
  The respiratory quotient will be measured by indirect calorimetry before and after consumption of a liquid mixed meal

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No